CLINICAL TRIAL: NCT03911258
Title: Epidemiology of the Nasal Flora at the Reference Center for Cystic Fibrosis of Queen Fabiola Children's University Hospital.
Acronym: FLONAMUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P2018/PNEUMO/FLONAMUC
Record Dates: First submitted 2019-03-04; First posted 2019-04-11 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal flora in CF patient (Experimental)
  Interventions: Procedure: nasopharyngeal swab versus nasal wash

INTERVENTIONS:
Procedure: nasopharyngeal swab versus nasal wash — The type of procedure will be determine according to patient collaboration

SUMMARY:
Cystic fibrosis (CF) is the most common autosomal recessive inherited genetic disorder in North America, Australia and Europe.

CF is due to cystic fibrosis transmembrane conductance regulator gene mutation (CFTR) coding for a chloride channel located at the apical membrane of epithelial cells. The most common mutation is the deletion of the amino acid phenylalanine at the codon 508 (ΔF508) affecting 70% of the patients.

The CFTR channel participates in the regulation of the volume and composition of exocrine secretions. At the level of the lungs, this results in a thickening of the mucus with a dysfunction of the mucociliary clearance promoting colonization of pathogenic microorganisms. Patients with cystic fibrosis therefore have a natural susceptibility to develop acute and then chronic respiratory infections, gradually leading to irreversible respiratory tract lesions called bronchiectasis. Different germs such as Haemophilus influenzae and Staphylococcus aureus colonize the airways early in life. The progression of the disease causes furthermore a colonization by opportunistic germs such as Pseudomonas aeruginosa and Burkholderia cepacia, which are associated with higher mortality.

Pulmonary exacerbation is a common complication of CF requiring administration of antibiotics. The choice of these antibiotics depends on the germs that the patient carries in his respiratory tract.

The type of sampling and the conditions under which they are taken are therefore very important. Sputum and oropharyngeal smear are used in adolescents and children respectively to collect respiratory secretions in clinical routine. The recent literature describes induced sputum, obtained after a physiotherapy session and a hypertonic serum aerosol, as superior to the oropharyngeal smear alone and equivalent to bronchoalveolar lavage for the evaluation of the microbiological profile of patients who cannot expectorate. However, this technique takes time and requires the presence of a physiotherapist.

Bronchoalveolar lavage is reserved for complex cases that do not respond to standard treatments.

Finally, the nasal flora appears to be involved in the colonization of the lower respiratory tract. Sinuses are described as reservoirs of germs that can induce a recolonization of the lungs despite eradication of the germ (for example after a pulmonary transplantation) .

To our knowledge, no study has investigated the involvement of nasal flora in the clinical course of children with CF.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients aged 0-20y followed in Cystic fibrosis at HUDERF
* For each participant, both parents or legally acceptable representative(s) must sign an informed consent form (ICF) indicating that they understand the purpose of, and procedures required for, the study and is willing to allow the child to participate in the study.
* Assent is also required of children capable of understanding the study (typically participants 7 years of age and older).

Exclusion Criteria:

Any clinical situation that prohibit the taking of samples as defined in this protocol:

* Severe respiratory distress
* An altered state of consciousness
* A pulmonary complication contrary to the realization of respiratory physiotherapy (pneumothorax, hemoptysis).

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
concordance between the microbiological results obtained by nasal lavage or swab and sputum in children | Day 1
  To see if there is any correlation in the cultures of pathogens present in the upper and lower respiratory tracts for any combination of samples taken

SECONDARY OUTCOMES:
Impact of upper respiratory microbial flora in the patient clinical course | Day 60
  To see if there is any correlation between the presence of pathogens in upper respiratory tract (URT) and the alteration of one or more clinical parameters at the time of sampling (BMI, FEV1, FVC, FEF25/75, Number of exacerbations)
Safety evaluation of the of the different methods of sampling | Day 1
  Type, frequency, severity and relationship between adverse events observed and sampling procedures performed.
Tolerance of the different methods of sampling | Day 1
  Pain / discomfort score induced by the set of sampling procedures measured by means of the "Visual Analogue Scale" (VAS) in children aged 5 or older. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (0) and 'pain as bad as it could be' (10). The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Tolerance of the different methods of sampling | Day 1
  Pain / discomfort score induced by the set of sampling procedures measured by means of the FLACC scale (Face, Legs, Activity, Cry, Consolability Scale) in children less than 5 years. FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2. The criteria evaluated are expression of the face, position of the legs, patient activity, type of cry, consolability
Tolerance of the different methods of sampling | Day 60
  Percentage of Drop-out for refusal of nasal sampling

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Beghin, MD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium